CLINICAL TRIAL: NCT00423917
Title: Phase II Trial of Fulvestrant and Bevacizumab in Patients With Metastatic Breast Cancer Previously Treated With an Aromatase Inhibitor
Brief Title: Fulvestrant and Bevacizumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0539; NCI-2009-00649 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000525570 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fulvestrant + bevacizumab (Experimental): Patients receive fulvestrant intramuscularly on day 1 and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, prior to every other course, and at the completion of study treatment.
  After completion of study treatment, patients are followed every 3-6 months for 5 years.
  Interventions: Biological: bevacizumab; Drug: fulvestrant

INTERVENTIONS:
Biological: bevacizumab
Drug: fulvestrant

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Fulvestrant and bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving fulvestrant together with bevacizumab may be an effective treatment for metastatic breast cancer.

PURPOSE: This phase II trial is studying how well giving fulvestrant together with bevacizumab works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy of fulvestrant and bevacizumab, in terms of 6-month progression-free survival (PFS), in patients with metastatic breast cancer previously treated with an aromatase inhibitor.

Secondary

* Assess the quality of life of patients treated with this regimen.
* Determine the adverse-event profile in these patients.
* Determine the PFS and overall survival of these patients.
* Determine the confirmed response rate, duration of response, time to treatment failure, and time to first cytotoxic agent in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive fulvestrant intramuscularly on day 1 and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, prior to every other course, and at the completion of study treatment.

After completion of study treatment, patients are followed every 3-6 months for 5 years.

PROJECTED ACCRUAL: A total of 51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Metastatic disease
* Must have received an aromatase inhibitor (e.g., letrozole, anastrozole, or exemestane) in an adjuvant or metastatic setting
* If tumor is HER2 positive (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization) the patient must have received ≥ 1 prior trastuzumab (Herceptin®)-containing regimen unless there is a contraindication to trastuzumab
* Measurable or nonmeasurable disease, including any of the following :

  * Bone metastasis
  * Pleural/pericardial effusion
  * Ascites
  * Inflammatory skin changes
* No microscopic residual disease only
* Enrolled on or refused enrollment on clinical trial NCCTG-N0392
* No evidence of active brain metastasis including leptomeningeal involvement

  * CNS metastasis controlled (i.e., at least 2 months of no symptoms or evidence of progression) by prior surgery and/or raditherapy are allowed
* Hormone receptor status:

  * Estrogen and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Male or female
* Female patients must be post-menopausal based on any 1 of the following criteria:

  * Age ≥ 60 years
  * Age ≥ 45 years with last menstrual period ≥ 12 months prior to study entry
  * Estradiol and follicle-stimulating hormone levels in postmenopausal range
  * History of bilateral oophorectomy
* ECOG performance status 0-2
* Life expectancy > 3 months
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* WBC ≥ 3,000 mg/dL
* Hemoglobin > 8 g/dL
* Absolute neutrophil count > 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Urine protein < 1+ OR < 1 g of protein by 24-hour urine collection

  * No nephrotic syndrome
* No uncontrolled hypertension (i.e., blood pressure [BP] > 160/90 mm Hg on ≥ 2 occasions at least 5 minutes apart)

  * Patients who have recently started or adjusted antihypertensive medications are eligible provided BP is < 140/90 mm Hg on any new regimen for ≥ 3 different observations in ≥ 14 days
* No clinically significant cardiac disease, including any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Unstable angina
  * Cardiac arrhythmias not well controlled with medication
  * Myocardial infarction within the past 12 months
* No arterial or venous thrombosis within the past 12 months
* No hemoptysis or gastrointestinal hemorrhage within the past 6 months
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 4 weeks
* No significant traumatic injury within the past 4 weeks
* No active, unresolved infection
* No history of hypertensive crisis or hypertensive encephalopathy
* No history of bleeding diathesis or uncontrolled coagulopathy
* No history of cerebrovascular accident, hemorrhage, or stroke
* No allergy or hypersensitivity to drug product excipients, murine antibodies, or agents chemically similar to study drugs
* No other malignancy within the past 3 years except for basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other serious medical condition that would preclude study therapy or compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior radiotherapy to a target lesion allowed provided there has been clear progression since radiotherapy was completed
* At least 4 weeks since prior radiotherapy

  * Single-dose radiation for palliation or to a nontarget lesion only allowed within the past 4 weeks
* No more than 1 prior chemotherapy regimen for metastatic disease
* No more than 2 prior endocrine (hormonal) therapy regimens in the neoadjuvant, adjuvant, or metastatic setting
* At least 4 weeks since prior major surgery or open biopsy
* At least 4 weeks since prior chemotherapy or immunologic therapy
* At least 2 weeks since prior and no concurrent use of any of the following agents:

  * Aspirin (daily low-dose [81 mg] aspirin allowed])
  * Thrombolytic agents
  * Anticoagulants (low-dose anticoagulation therapy to maintain patency of a vascular access device is allowed)
* No concurrent treatment in another clinical study with investigational procedures or investigational therapies
* No other concurrent anticancer therapy, including chemotherapy, biologic agents, or radiotherapy
* No routine use of granulocyte colony-stimulating factors during course 1
* No concurrent oprelvekin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2017-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Tan, MD, FACP, Study Chair — Mayo Clinic
Locations (205):
- United States (205):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Tan WW, Dueck AC, Flynn P, Steen P, Anderson D, Rowland K, Northfelt D, Perez EA. N0539 phase II trial of fulvestrant and bevacizumab in patients with metastatic breast cancer previously treated with an aromatase inhibitor: a North Central Cancer Treatment Group (now Alliance) trial. Ann Oncol. 2013 Oct;24(10):2548-2554. doi: 10.1093/annonc/mdt213. Epub 2013 Jun 24. PMID 23798616

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant + Bevacizumab: Patients receive Fulvestrant 250 mg intramuscularly every 28 days and Bevacizumab 10mg/kg intravenously with a rate-regulating device on days 1 and 15. Loading dose of fulvestrant for the first cycle will consist of an extra 250 mg on day 1 (for total of 500 mg Cycle 1, Day 1). The initial bevacizumab dose will be delivered over 90 minutes. If the first infusion is tolerated without infusion-associated adverse events (fever and/or chills), the second infusion may be delivered over 60 minutes. If the 60-minute infusion is well-tolerated, all subsequent infusions may be delivered over 30 minutes.Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Fulvestrant + Bevacizumab
Started | 36
Completed | 33
Not Completed | 3
Not completed — Cancel | 2
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 65 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Six-month Progression-free Survival (PFS) Rate at 6 Months
Description: The primary endpoint of this trial is the 6-month progression-free survival rate. A patient is considered to be a 6-month progression-free survivor if the patient is on study treatment 6 months from registration without a documentation of disease progression. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Additionally, if some patients are lost to follow-up not having been observed for at least 6 months, an estimate and 95% confidence interval for the 6-month progression-free survival rate incorporating censoring will be computed using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
percentage of patients | 39 [23 to 58]

2. Secondary Outcome: Progression Free Survival
Description: Time to disease progression is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression 1 day post-registration. The distribution of time to progression will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
months | 6.2 [3.6 to 10.1]

3. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier (1958).
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
months | 26.9 [12.5 to 36.2]

4. Secondary Outcome: Quality of Life, as Measured by the Largest Mean Change in LASA Overall QOL and Physical Well-being Items
Description: Quality of life (QOL) assessment will be a secondary exploratory component of this trial. QOL of patients was measure using the 6-item Linear Analogue Self-Assessment (LASA).The LASA consists of six single-item numeric analog scales measuring overall QOL; mental, physical, emotional, and spiritual well-being; and level of activity each on a scale of 0 ('As bad as it can be') to 10 ('As good as it can be') during the past week. Items were transformed to a 0 (worst QOL or well-being) to 100 (best QOL or well-being) scale for statistical analysis. Mean change from baseline of the largest mean change in overall QOL and physical well-being are reported below.
Time Frame: Up to 5 years
Measure: Mean (Standard Deviation); unit: mean change in LASA QOL scaled score
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
mean change in LASA QOL scaled score
  Overall Quality of Life | -5.0 (15.0)
  Physical Well-Being | -6.8 (14.9)

5. Secondary Outcome: Objective Response Rate as Measured by RECIST Criteria in Patients With Measurable Disease
Description: A confirmed response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. The confirmed response rate will be estimated by the number of confirmed responses in evaluable patients with measurable disease divided by the total number of evaluable patients with measurable disease. The appropriate confidence interval will be calculated. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 18
percentage of patients | 22 [6 to 22]

6. Secondary Outcome: Time to First Cytotoxic Agent
Description: Time to first dose of a cytotoxic agent is defined to be the time from the date of registration to the date at which a patient recieves the first dose of a cytotoxic agent. The distribution of time to first dose of a cytotoxic agent will be estimated using the method of Kaplan-Meier (1958).
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 33
months | 9.9 [6.2 to 19.5]

7. Secondary Outcome: Duration of Response/Time to Disease Progression in Patients With Measurable Disease
Description: Duration of response is defined for all evaluable patients with measurable disease who have achieved a confirmed response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented. If a patient dies subsequent to the confirmed response without a documentation of disease progression, the patient will be considered to have had disease progression at the time of their death. In the case of a patient failing to return for evaluations before a documentation of disease progression, the patient will be censored for progression on the date of last evaluation. The distribution of duration of response will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 5 years
Population: Evaluable patients with measurable disease who experienced a confirmed response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant + Bevacizumab
Number analyzed (Participants) | 4
months | 11.9 [3.7 to NA] — The upper limit of the 95% confidence interval for Duration of Response in Patients with Measurable Disease who experienced a confirmed response was not reached.

ADVERSE EVENTS:
Time Frame: Adverse events are assessed 14 days prior to registration, prior to each treatment cycle, and at the end of treatment.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized until March 31, 2011. CTCAE version 4.0 will be utilized for expedited adverse event reporting only, beginning April 1, 2011. All appropriate treatment areas should have access to a copy of the CTCAE v4.0.
Arm/Group | Fulvestrant + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 4/33
Other Adverse Events (participants affected / at risk) | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Bevacizumab (N=33)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Bevacizumab (N=33)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (7)
Left ventricular failure (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (47)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (10)
Nausea (Gastrointestinal disorders) | 15 (43)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (20)
Vomiting (Gastrointestinal disorders) | 4 (8)
Fatigue (General disorders) | 6 (14)
Fever (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 13 (48)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 3 (16)
Creatinine increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (13)
Memory impairment (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 11 (57)
Renal failure (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (45)
Hot flashes (Vascular disorders) | 2 (4)
Hypertension (Vascular disorders) | 11 (42)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes